CLINICAL TRIAL: NCT06033768
Title: Neurological and Psychological Assessment of Neurocutaneous Syndromes in Upper Egypt Children
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamad, doctor, Assiut University
Other Study IDs: Ncs compilications
Record Dates: First submitted 2023-09-03; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Neurocutaneous Syndromes
MeSH Terms: conditions — Neurocutaneous Syndromes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Evaluation of neurological and psychological complications in children diagnosed as neurocutaneous syndromes in upper Egypt

DETAILED DESCRIPTION:
Neurocutaneous syndromes (NCS) are heterogeneous group of disorders characterized by abnormalities of both the integument and central nervous system. Most of the disorders of NCS are inherited as autosomal dominant conditions and originated from a defect in differentiation of the primitive ectoderm.NCS include Neurofibromatosis1 (NF1), Tuberous Sclerosis (TS), Sturge Weber Syndrome (SWS), von Hippel-Lindau disease (VHL), Pascual-Castroviejo type II syndrome (PHACE syndrome), Ataxia telangiectasia (AT),Linear Nevus Syndrome (LNS), hypo melanosis of Ito and Incontenintia Pigmenti(IP), Xeroderma pigmentosa (XP). Among them the most common disorders areNF, TS complex and SWS. These lifelong disorders generally present during infancy and early childhood..These disorders are characterized clinically by neurological manifestations as convulsions, mental retardation and learning disabilities.

Tuberous sclerosis complex (TSC) is an autosomal dominant genetic disorder that is diagnosed from birth to adulthood.TSC is characterized by growth of non-malignant hamartoma in various organs throughout the body.

The majority of individuals with Tuberous sclerosis have mutations in either the TSC1 orTSC2 genes.

Most common manifestations of Tuberous sclerosis are multiple type of seizures and various organ involvement.

Epilepsy is very common in people living with Tuberous Sclerosis Complex (TSC), with around 8 in every 10 children with Tuberous Sclerosis also experiencing epilepsy.Epilepsy in Tuberous Sclerosis often begins during the first year of life and,in most cases, in the first month. At this time the most common types of seizures are partial motor seizures and infantile spasms.

Many of the multi-dimensional problems experienced by patients with Tuberous sclerosis changeover time, substantially affecting quality of life. Thus, an overall understanding of physical, cognitive, and mental health is necessary to ensure continuous and systematic management of symptoms in this population.

Among the psychiatric problems associated with Tuberous sclerosis, autism spectrum disorder (ASD) is the most common, affecting up to 61 % of patients However, its severity is not frequently reported, and the risk factors for autism spectrum disorder in the Tuberous sclerosis population are still controversial.

Numis et al. followed 103 patients with Tuberous sclerosis, and 40% had concurrent autism .

The neurocognitive panel of the 2012 International Tuberous sclerosis Consensus Conference recommended that individuals with Tuberous sclerosis should be screened for comorbid conditions once per year.In 2015, DeVries et al. proposed the Tuberous Sclerosis-AssociatedNeuropsychiatric Disorders (TAND) checklist. Neurofibromatosis 1 (NF1) is an umbrella term for 3 genetically distinct disorders:NF1, NF2, and Schwannomatosis. They have a common tendency toward development of tumors of the nerve sheath, but the specific manifestations are distinct and the conditions result from variants indifferent genes. NF1 is the commonest neurofibromatosis and the most likely to present in childhood. Café- au-lait macules are the pathognomonic cutaneous manifestations of NF1 thatpresent at birth but often gradually appear in the first few postnatal months .

The most common complications of NF1 are cognitive and behavioral deficits,Upto 80% of children with NF1 experience cognitive and behavioral difficulties involving different domains. Parents often report poor performance in reading,written work, spelling, organizational skills, and mathematics. In addition,approximately 38% of affected children have attention-deficit/hyperactivity disorder (ADHD),and some studies have reported that 29% of children with NF1have autism spectrum disorder (ASD ) Ataxia-telangiectasia is a multisystem disorder characterized by progressive deterioration of neurologic function, ocular and cutaneous telangiectasia, cerebellar ataxia and variable immunodeficiency .

Ataxia telangiectasia is an autosomal recessive neurodegenerative disorder that is characterized by progressive cerebellar atrophy and ataxia,radio sensitivity, immune deficiency and tendency to develop lymphoreticular malignancies. The disorder is relatively rare, with an incidence of 1:40000 to 1:100 000. It is the secondmost frequent cause of recessive ataxia in childhood after Freidreich ataxia, but the most frequent in children with onset of ataxia within the first years of life .

Sturge-weber syndrome is defined as the occurrence of port-wine stain on the face associated with leptomeningeal angiomatosis that can lead to seizures, stroke and glaucoma. The port-wine stain can occur without leptomeningeal involvement and leptomeningeal involvement can occur without the port-wine stain .

The main neurological complication of Sturge Weber Syndrome are seizures (75% to 90%), slowly progressive hemi paresis (25% to 60%), migraine-like vascular headaches (30% to 45%), delayed neuropsychological development (50%to 60%), episodes similar to cerebro-vascular events, with acute transient hemiplegia, visual field defects, and behavioral problems.

Xeroderma pigmentosum is a rare autosomal recessive genodermatosis due to mutations in nucleotide excision repair. The condition characteristicallydemonstrates severe photosensitivity, skin pigmentary changes, malignant tumordevelopment, and occasionally progressive neurologic degeneration. The disease affects about 1 per million in the United States, and the incidence in Japan ismuch higher at 45 per million.

Von Hippel-Lindau disease is named after Eugen Von Hippel, a German ophthalmologist and Arvid Lindau, a Swedish pathologist. In 1904 Von Hippel first described angiomas in the eye, while Lindau described angiomas of the cerebellum and spine in 1927. As a result, the term "VHLDisease" was first used in 1936 and gained acceptance and became established in the medical literature from the 1970. Von Hippel-Lindau disease is characterized by hemangioblastomas of the brain, spinal cord, andretina. Renal cysts and clear cell renal cell carcinoma,Pheochromocytoma, pancreatic cysts, and neuroendocrine tumors,Endolymphatic sac tumors and epididymal and broad ligament cysts.

PHACE syndrome is a neurocutaneous condition in which extensive or segmental infantile hemangioma (IH), usually on the face, scalp, or cervical region,can be associated with posterior fossa malformations, arterial abnormalities [primarily inthe CNS], coarctation of the aorta, cardiac defects, and ocular abnormalities.

Incontentia Pigmenti is a rare X-linked dominant disorder that affects the skin,teeth, eyes, central nervous system, and skeletal system . As an X-linked trait, it is usually lethal to males, hence the preponderance of females with this condition. In fact, females represent about 98% of babies born with Incontentia Pigmenti. Incontentia Pigmenti is a multisystem disorder with prominent features of mosaicism or cutaneous patterns that connote an individual comprised of two or more different cell lines.

Hypomelanosis of Ito is a pigmentary mosaicism characterized by a clone of skin cells with decreased ability to produce pigment. The clinical patterns characterized by hypo pigmented streaks and whorls running along the lines of Blaschko, characteristically involving more than two body segments.

Cerebral malformations may occur, and visual impairment may be cortical in nature with Hypomelanosis of Ito.

The Diagnostic and Statistical Manual of Mental Disorders (DSM) is the handbook widely used by clinicians and psychiatrists in the United States to diagnose psychiatric illnesses. Published by the American Psychiatric Association (APA), the DSM covers all categories of mental health disorders for both adults and children. It contains descriptions, symptoms, and other criteria necessary for diagnosing mental health disorders. It also contains statistics concerning who is most affected by different types of illnesses, the typical age of onset, the development and course of the disorders, risks and prognostic factors, and other related diagnostic issues.

One of the most trouble some aspects in the exploration of the affective and behavioraldysregulation is the difficulty of reliable and cost-effective diagnostic measures. The Child Behavior Checklist (CBCL), one of the most frequently used instruments for assessment of developmental psychopathology.

In TSC the term TAND (Tuberous Sclerosis Associated Neuropsychiatric Disorders) is used to capture the multidimensional biopsychosocial difficulties of the disease.

A specific TAND Checklist has been developed to assess Behavioral, Psychiatric, Intellectual, Academic, Neuropsychological and Psychosocial areas .

To date, no psychosocial disease-specific screening tool has been developed toassess other nurocutaneous syndromes patients .

ELIGIBILITY:
Inclusion Criteria:

- All children with sign and symptoms of neurocutneous syndromes.

Exclusion Criteria:

* Children with pigmentary and neurological disorders other than neurocutneous syndromes.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: his study will be carried out in outpatient clinic and inpatient department in Assiut University Children's Hospital .
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
epilepsy | baseline
  prevalence of epilepsy in children with neurocutaneous syndromes
autism spectrum | baseline
  prevalence of autism spectrum in children with neurocutaneous syndromes
attention deficit hyperactivity syndrome | baseline
  prevalence of attention deficit hyperactivity syndrome in children with neurocutaneous syndromes
depression | bsaeline
  prevalence of depression in children with neurocutaneous syndromes